CLINICAL TRIAL: NCT05155033
Title: Phase II Trial of Combination Anti-PD-1 and Aldesleukin for Metastatic Melanoma and Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000354; 000354-C
Record Dates: First submitted 2021-12-10; First posted 2021-12-13 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01-20

CONDITIONS: Metastatic Melanoma; Advanced Locoregional Melanoma; Metastatic Renal Cell Carcinoma; Clear Cell Histology
Keywords: Immunotherapy; Monoclonal Antibody
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell | interventions — pembrolizumab; aldesleukin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 - Pembro and IL-2 (Experimental): Course 1: pembrolizumab (200 mg IV) on Day 1 of each cycle with aldesleukin (600,000 IU/kg intravenous bolus every eight hours) continuing for up to 4 days (maximum 10 doses) for 2 cycles (each 21 days). Course 2: pembrolizumab (200 mg IV) on Day 1 of each cycle for 2 cycles (each 21 days).
  Interventions: Drug: Pembrolizumab; Drug: Aldesleukin

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg IV over approximately 30 minutes on Day 1 of cycles 1 and 2 during Courses 1 and 2.
Drug: Aldesleukin — Aldesleukin (IL-2) administration [600,000 IU/kg IV bolus every 8 hours continuing for up to 4 days (maximum 10 doses)] starting on Day 1 of cycles 1 and 2 during Course 1.

SUMMARY:
Background:

Aldesleukin is used to treat metastatic or advanced melanoma and renal cell carcinoma. Pembrolizumab is used to treat many cancers including melanoma. Researchers want to see if these drugs can be used together to produce better results in people with these types of cancer.

Objective:

To learn if the combination of pembrolizumab and aldesleukin can be used to treat metastatic or advanced melanoma and renal cell cancer.

Eligibility:

Adults aged 18 years or older who have metastatic or advanced melanoma or renal cell carcinoma.

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Electrocardiogram
* Blood and urine tests
* Ability to perform tasks of daily living
* Imaging scans (CT, MRI, PET, and/or X-rays). They may get a contrast agent to enhance the images.
* Photographs, if needed

Some of these tests will be repeated during the study.

Participants will receive the study drugs by IV (a plastic tube that is put into a vein) for 4 days. A second cycle of treatment will be given 21 days later. They will stay in the hospital for each of the cycles in the first course of treatment. After 2 months, their cancer will be evaluated. They may receive a second course of pembrolizumab alone on Days 1 and 21. They will not have to stay in the hospital for this course.

About 30 days after treatment ends, participants will have a safety follow-up visit. Then they will have visits every 3 months for up to 1 year, and then every 6 months for up to 4 years. Follow-up can also be done by phone, email, and mail. If their cancer gets worse, they will stop having visits.

Participation will last for 5 years.

DETAILED DESCRIPTION:
Background:

High-dose interleukin-2 was approved by the FDA for the treatment of metastatic melanoma and renal cell carcinoma, with overall response rates of 15-16%. Complete regression of disease was seen in 6-7% of participants with many long-term durable responses. The regimen has not been widely adopted due to complexities in management and the development of alternative effective therapies, such as monoclonal antibodies targeting immune checkpoints (ipilimumab, pembrolizumab, nivolumab) or small molecule inhibitors.

Pembrolizumab was approved by the FDA for the treatment of metastatic melanoma based on a series of studies demonstrating objective response rates from 21-34%. There remains a considerable population of participants with disease that never responded to treatment, in addition to participants with short durations of response prior to recurrence.

There has been limited clinical investigation of the combination of interleukin-2 and pembrolizumab. The hypothesis under investigation is that non-specific activation of the immune system with both positive stimulation (aldesleukin) and release of negative regulation (pembrolizumab) may have meaningful clinical impact for participants with limited therapeutic options.

Objectives:

Primary:

To determine the objective response rate as determined by RECIST 1.1 criteria to combined aldesleukin and pembrolizumab in participants with advanced melanoma refractory to anti-PD-1 therapy and treatment-refractory metastatic renal cell carcinoma

Secondary:

To determine progression free survival with the combined regimen

To determine the toxicity profile of this treatment regimen

To determine the objective response rate as determined by RECIST 1.1 criteria to combined aldesleukin and pembrolizumab in participants with treatment-na(SqrRoot) ve advanced melanoma

Exploratory:

To evaluate clinical and laboratory correlates of response

To perform immunologic correlative studies of peripheral blood, tumor, and/or tumor infiltrating lymphocytes including but not limited to phenotype and functional analysis of longitudinal samples

Eligibility:

Participants must be/have:

Age >= 18 years of age.

ECOG performance status of 0 or 1.

Expected survival of greater than 6 months.

Histologically or cytologically confirmed melanoma or renal cell cancer, as follows:

Cohort 1: Metastatic melanoma or advanced locoregional melanoma not amenable to curative surgical resection and refractory to anti-PD-1 therapy.

Cohort 2: Metastatic renal cell carcinoma (clear cell histology) refractory to at least one line of PD1/PDL1 based therapy.

Cohort 3: Metastatic or advanced locoregional melanoma not amenable to curative surgical resection na(SqrRoot) ve to anti-PD-1 therapy.

No allergies or hypersensitivity to high-dose aldesleukin or pembrolizumab administration.

No concurrent major medical illnesses or any form of immunodeficiency.

No history of Grade 3/4 immune-related adverse events affecting major organ systems associated with the administration of single agent pembrolizumab or nivolumab.

Design:

Study treatment will be given in two courses. A course shall consist of two cycles (each 21 days) of treatment. Cycles in Course 1 shall consist of pembrolizumab (200 mg IV) infusion on the morning of Day 1 with aldesleukin (IL-2) administration (600,000 IU/kg intravenous bolus every eight hours) to begin later that day. IL-2 will be administered to tolerance or to a maximum of 10 doses.

A second cycle of treatment will begin during Week 4 (Day 22-28).

Approximately two months from the beginning of therapy, participants will be evaluated for response including physical exam, clinical laboratory testing, and cross-sectional imaging.

Participants that do not demonstrate progressive disease will receive a second course of pembrolizumab alone, if clinically appropriate.

Participants with stable disease will be monitored until disease progression (every 3 months x 3) up to one year.

Participants with an objective response will be monitored until disease progression (every 3 months x 3, every 6 months x 8) up to five years.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically or cytologically confirmed cancer that falls into one of three cohorts: (1) metastatic melanoma or advanced locoregional melanoma not amenable to curative surgical resection and refractory to anti-PD-1 therapy; (2) metastatic renal cell carcinoma (clear cell histology) refractory to at least one line of PD1/PDL1 based therapy; (3) metastatic or advanced locoregional melanoma not amenable to curative surgical resection and naive to anti-PD-1 therapy.
* Participants must have measurable disease (per RECIST v1.1 criteria), metastatic melanoma or renal cell cancer.
* Age >=18 years of age.
* Clinical performance status of ECOG 0 or 1.
* Willing to practice birth control from the time of enrollment on this study and for four months after treatment.
* Must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
* Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Participants who are HIV seropositive may have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
* Seronegative for hepatitis B antigen and for hepatitis C antibody. If hepatitis C antibody test is positive, then participant must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
* Participants must have adequate organ and marrow function as defined below:

  * ANC > 1000/mm^3 without the support of filgrastim
  * WBC >= 3000/mm^3
  * Platelet count >= 100,000/mm^3
  * Hemoglobin > 8.0 g/d (Subject may be transfused to reach this cut-off)
  * Serum ALT/AST <= 5.0 x ULN
  * Serum creatinine <= 1.6 mg/dL
  * Total bilirubin <= 2.0 mg/dL, except in participants with Gilbert s Syndrome, who must have a total bilirubin < 3.0 mg/dL.
* More than four weeks must have elapsed since completion of any prior systemic therapy at the time of enrollment.

Note: Participant may have undergone minor surgical procedures or limited field radiotherapy within the four weeks prior to enrollment, as long as related major organ toxicities have recovered to <= grade 1.

* Ability of subject to understand and the willingness to sign a written informed consent document.
* Willing to sign a Durable Power of Attorney Form.
* Subject must be co-enrolled on protocol 03-C-0277

EXCLUSION CRITERIA:

* Participant is nursing because of the potentially dangerous effects of the treatment on the fetus or infant.
* Concurrent systemic steroid therapy.
* Active systemic infections requiring anti-infective treatment, coagulation disorders, or any other active or uncompensated major medical illnesses.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and AIDS).
* History of major organ autoimmune disease.
* Grade 3 or 4 major organ irAEs following treatment with anti-PD-1/PD-L1 monotherapy, including but not limited to myocarditis, pneumonitis, colitis, and hepatotoxicity.
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Participants who have decreased immune-competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
* History of severe immediate hypersensitivity reaction to pembrolizumab or aldesleukin.
* History of coronary revascularization or ischemic symptoms.
* For select participants with a clinical history prompting cardiac evaluation: last known LVEF <= 45%.
* For select participants with a clinical history prompting pulmonary evaluation: known FEV1 <= 50%.
* Participant is receiving any other investigational agents.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2031-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Response rate in treatment refractory disease | 8 weeks after Course 1 Cycle 1 then after Course 2, every 3 months x 3 (up to one year), every 6 months x 8 (up to five years)
  Determine the rate of objective response (using RECIST v1.1 criteria)

SECONDARY OUTCOMES:
Progression Free Survival | Every 2-6 months for up to 5 years
  Elapsed duration from enrollment to progression of disease
Response rate in treatment naive melanoma | 8 weeks after Course 1 Cycle 1 then after Course 2, every 3 months x 3 (up to one year), every 6 months x 8 (up to five years)
  Determine the rate of objective response (using RECIST v1.1 criteria)
Safety and tolerance | First dose through 30 days after last treatment
  Using standard CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L Goff, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.@@@@@@All collected IPD will be shared with collaborators under the terms of collaborative agreements
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000354-C.html